CLINICAL TRIAL: NCT02473614
Title: To Determine the Therapeutic Effect of the Music Glove and Conventional Hand Exercises
Brief Title: Efficacy Study of the Music Glove Patients With Spinal Cord Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Kelli Sharp, Assistant Professor at the Department of Dance, University of California, Irvine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2R44HD074331-02 [2008-6432]; 2R44HD074331-02 (NIH)
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music Glove (Experimental): Music Glove is a glove with sensors attached to the tips of all 5 fingers. The glove is connected to a software musical program like guitar hero. Participants will follow the rhythm or musical notes of the songs and move their fingers accordingly. Participants are reinforced with biofeedback that includes visual and auditory cues when the correct sequences are achieved.
  Interventions: Device: Music Glove
- Conventional Hand Exercise Program (Active Comparator): Conventional Hand Exercise Program includes range of motion exercises, strengthening exercises, coordinating exercises of the hand and fingers. This exercise program is designed by an occupational therapist and is a general exercise program that a stroke patient will receive when he/she is being discharged from the hospital.
  Interventions: Other: Conventional Hand Exercise Program

INTERVENTIONS:
Device: Music Glove — Participants will exercise at home using the music glove for 3 times a week for 3 weeks with a minimum of 3 hours per week.
  Arms: Music Glove
Other: Conventional Hand Exercise Program — Participants will exercise at home using the hand exercise program designed by an occupational therapist for 3 times a week for 3 weeks with a minimum of 3 hours per week.
  Arms: Conventional Hand Exercise Program

SUMMARY:
Investigators are trying to determine the therapeutic effect of the music glove and conventional hand exercise program to patients with spinal cord injuries. All participants will be randomized into two groups: AB and BA. They will all exercise at least 3 times a week for 3 weeks with minimum of 3 hours of exercise time per week. Participants will receive the other intervention at their 3 week post-therapy follow-up visits. Clinical evaluations will be performed at baseline 1 and 2 (3 to 10 days apart), post-therapy after the first intervention, 3-week post-therapy follow up, post-therapy after the second intervention, and 3-week post-second intervention follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* History of spinal cord injury affecting the arm and hand functions, at least 6 months prior to enrollment
* Upper extremity weakness as measured on a standard clinical scale
* No active major psychiatric problems, or neurological/orthopedic problems affecting the training upper extremity
* No active major neurological disease other than the spinal cord injury
* Absence of pain in the affected upper extremity

Exclusion Criteria:

* Severe tone at the affected upper extremity as measured on a standard clinical scale
* Severe sensory/proprioception deficit at the affected upper extremity as measured on a standard clinical scale
* Difficulty in understanding or complying with instructions given by the experimenter
* Inability to perform the experimental task that will be studied
* Increased pain with movement of the training upper extremity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Sharp, DPT, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

REFERENCES:
- [Derived] Sanders Q, Chan V, Augsburger R, Cramer SC, Reinkensmeyer DJ, Sharp K. Feasibility of home hand rehabilitation using musicglove after chronic spinal cord injury. Spinal Cord Ser Cases. 2022 Nov 9;8(1):86. doi: 10.1038/s41394-022-00552-4. PMID 36347833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 subjects were screened for eligibility
Pre-assignment Details: 11 of the 34 participants were randomized.
Groups:
- Music Glove First, Then Conventional Hand Exercise Program: Participants first participated in Music Glove therapy intervention for 3 times a week for 3 weeks with a minimum of 3 hours per week. After a washout period of 3 weeks, they participated in a conventional hand therapy program for 3 weeks with a minimum of 3 hours per week.
- Conventional Hand Exercise Program First, Then Music Glove: Participants first participated in conventional hand therapy for 3 times a week for 3 weeks with a minimum of 3 hours per week. After a washout period of 3 weeks, then they participated in the Music Glove therapy intervention for 3 weeks with a minimum of 3 hours per week.
Period: First Intervention (3 Weeks)
Arm/Group | Music Glove First, Then Conventional Hand Exercise Program | Conventional Hand Exercise Program First, Then Music Glove
Started | 6 | 5
Completed | 5 | 5
Not Completed | 1 | 0
Not completed — Job duties/lack of transportation | 1 | 0
Period: Wash Out Period (3 Weeks)
Arm/Group | Music Glove First, Then Conventional Hand Exercise Program | Conventional Hand Exercise Program First, Then Music Glove
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention (3 Weeks)
Arm/Group | Music Glove First, Then Conventional Hand Exercise Program | Conventional Hand Exercise Program First, Then Music Glove
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to participate in Music Glove or Conventional Hand Exercise Program for 3 weeks, then after a three-week washout period they participated in either Music Glove or Conventional Hand Exercise Program for 3 weeks.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Box and Blocks Test
Description: We compared the change of Box and Blocks Test (BBT) scores from baseline evaluation to the end of 3-week of therapy, and from 1-month post first intervention to the end of the second 3-week therapy. Participants are instructed to move as many blocks as possible, one at a time, from one compartment in a box to a second compartment over a divider for a period of 60 seconds; each block that is moved is counted, and multiple blocks moved at the same time are counted as a single block. The higher scores indicate better outcomes.
Time Frame: Baseline, EOT 1st Intervention, 1 month post 1 intervention, EOT 2nd Intervention, and 1 month post 2nd Intervention.
Measure: Mean (Standard Deviation); unit: blocks
Arm/Group | Music Glove First, Then Conventional Hand Exercise Program | Conventional Hand Exercise Program First, Then Music Glove
Number analyzed (Participants) | 5 | 5
blocks
  Baseline | 40.6 (1.7) | 40 (18.0)
  EOT 1st Intervention (3 weeks) | 44.8 (7.0) | 39.0 (19.6)
  1Month Post 1st Intervention | 46.4 (1.7) | 41.0 (22.2)
  EOT 2nd Intervention | 43.0 (4.8) | 43.2 (20.9)
  1-month Post 2nd Intervention | 46.6 (6.1) | 40.4 (22.0)

2. Secondary Outcome: Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP)
Description: We used the GRASSP to capture information on upper limb impairment from the SCI population through three domains: Strength, Sensibility, and Prehension. We focused on the Prehension section of the test. The prehension ability domain consists of three different tasks 1) Cylindrical Grasp, 2) Lateral Key Pinch, & 3) Tip to Tip Pinch and one can score 0-4 for each task for a total of 12 points for this section. The prehension performance domain consists of 1) pour water from a bottle, 2) open jars, 3) pick up & turn a key, 4) transfer 9 pegs board to board, 5) pick up 4 coins & place in the slot, 6) screw 4 nuts onto bolts and one can score 0-5 for each task for a total of 30 points. The score for each domain of the prehension test is totaled for each of the upper extremities with ranges from 0 to 42. The higher scores indicate better functional outcomes.
Time Frame: Baseline, EOT 1st Intervention, 1 month post 1 intervention, EOT 2nd Intervention, and 1 month post 2nd Intervention.
Measure: Mean (Standard Deviation); unit: points
Groups:
- Conventional Hand Exercise Program: Participants first participated in conventional hand therapy for 3 times a week for 3 weeks with a minimum of 3 hours per week. After a washout period of 3 weeks, then they participated in the Music Glove therapy intervention for 3 weeks with a minimum of 3 hours per week.
Arm/Group | Music Glove First, Then Conventional Hand Exercise Program | Conventional Hand Exercise Program
Number analyzed (Participants) | 5 | 5
points
  Baseline | 18.6 (3.0) | 18.6 (6.1)
  EOT 1st Intervention | 20.0 (5.1) | 19.0 (6.4)
  1-month post 1st Intervention | 19.6 (4.2) | 20.6 (4.4)
  EOT 2nd Intervention | 20.2 (3.8) | 21.1 (4.8)
  1-month post 2nd Intervention | 20.8 (4.1) | 20.2 (5.7)

ADVERSE EVENTS:
Time Frame: Through study completion an average of 12 weeks.
Groups:
- Music Glove: Participants participated in Music Glove therapy intervention 3 times a week for 3 weeks with a minimum of 3 hours per week.
- Conventional Hand Exercise Program: Participants participated in conventional hand therapy 3 times a week for 3 weeks with a minimum of 3 hours per week.
Arm/Group | Music Glove | Conventional Hand Exercise Program
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No